CLINICAL TRIAL: NCT05832138
Title: ONLOOP Trial: Evaluating a New Surveillance and Support System for Survivors of Childhood Cancer in Ontario
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Women's College Hospital (Other); Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Paul Nathan, Staff Oncologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 4152
Record Dates: First submitted 2023-04-14; First posted 2023-04-27 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Survivorship; Cancer; Heart Diseases; Secondary Cancer; Colorectal Cancer; Breast Cancer
Keywords: Surveillance; Guideline-recommended surveillance; Implementation science; Reminder system; Intervention
MeSH Terms: conditions — Neoplasms; Heart Diseases; Neoplasms, Second Primary; Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Usual care plus ONLOOP program materials:
  1. Study invitation letter and invitation reminder 5 weeks later
  2. For those who sign up: receipt of a personalized health toolkit and then a screening reminder 6 months later
  3. Optional: Engagement of primary care provider through an introductory letter and then a reminder letter sent 6 months later
  Interventions: Behavioral: ONLOOP program
- Delayed Intervention (Other): Usual care plus delayed ONLOOP:
  Survivors will receive usual care for 13 months after study invitation packages are mailed out to the intervention arm. At that point, survivors in this group will also receive the study invitation package.
  Interventions: Behavioral: ONLOOP program

INTERVENTIONS:
Behavioral: ONLOOP program — Participants will receive ONLOOP program intervention materials: a study invitation letter, personalized health information, and a reminder to complete their guideline-recommended surveillance test(s)

SUMMARY:
The treatments that aim to cure cancer in children can lead to "late effects" such as second cancers and heart disease. Screening tests can help find late effects, but most adult survivors of childhood cancer do not complete these tests. These survivors are at risk for harm that can be prevented.

The investigators have developed a program called ONLOOP to remind survivors in Ontario, Canada to get the screening tests they need. ONLOOP reminds survivors who are at higher risk for heart disease, breast cancer, and/or colorectal cancer to complete their echocardiograms, mammograms and breast MRIs, and/or colonoscopies.

The goal of this clinical trial is to find out how well ONLOOP helps adult survivors of childhood cancer complete their screening tests. The investigators also want to see if it could be turned into a long-term program in Ontario. Eligible survivors will be randomly assigned to either receive intervention materials or continue with usual care for 13 months before receiving intervention materials.

The intervention includes usual care plus these ONLOOP materials:

1. Study invitation letter and invitation reminder
2. Those who sign up for ONLOOP will receive personalized health information and a screening reminder. Survivors will receive information about:

   1. their cancer treatment
   2. their risk(s) for late effects
   3. the screening tests they should do
3. Participants have the option to provide their family doctor's or nurse practitioner's contact information. For those who consent, the study team will send their family doctor or nurse practitioner a letter with details about their cancer diagnosis and treatment. The letter will also remind them to talk to their patient about their health and screening test(s) needed.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of childhood cancer who are currently aged 18 and older
* Diagnosed with cancer before age 18 between 1986-2017
* At least 5 years from most recent childhood cancer event (latest of primary diagnosis, relapse, or second cancer before age 18)
* Treated at one of Ontario's five specialized childhood cancer programs
* Received radiation and/or anthracycline treatment that increased the survivor's risk of cardiomyopathy, breast cancer, and/or colorectal cancer
* Overdue for guideline-recommended surveillance by ≥6 months (mammogram and breast MRI, colonoscopy, and/or echocardiogram)

Exclusion Criteria:

* Was not diagnosed or was not fully treated at one of Ontario's five pediatric cancer centres
* Developed a second cancer or relapse of their primary cancer after age 18
* Not currently living in Ontario or address deemed ineligible by Ontario Health
* Opted out of a similar Ontario Health program (eg, the Ontario Breast Screening Program)
* Previously opted out of receiving invitations for Ontario Health research studies or similar communications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Completion of guideline-recommended surveillance tests | 12 months
  Proportion of survivors who complete one or more of the guideline-recommended cardiac, breast or colon surveillance tests (echocardiography, mammogram and breast MRI, colonoscopy) during the 12 months after study cohort randomization

SECONDARY OUTCOMES:
Completion of guideline-recommended surveillance tests | 24 months
  Proportion of survivors who complete one or more of the guideline-recommended cardiac, breast or colon surveillance tests (echocardiography, mammogram and breast MRI, colonoscopy) during the 24 months after study cohort randomization
Completion of each type of surveillance test | 12 months, 24 months
  Proportion of survivors who complete each type of surveillance test (among those eligible for the test)
Completion of all guideline-recommended surveillance tests | 12 months, 24 months
  Proportion of survivors who are fully up-to-date according to surveillance guidelines
Visits to primary care professionals and cancer specialists | 12 months, 24 months
  Number of outpatient visits to primary care professionals and to cancer specialists
Use of other healthcare services | 12 months, 24 months
  Rates of emergency department visits and/or hospitalizations to understand impact on health system resources

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nathan, MD, MSc, Principal Investigator — The Hospital for Sick Children; Noah Ivers, MD, PhD, Principal Investigator — Women's College Hospital

REFERENCES:
- [Derived] Shuldiner J, Lam E, Shah N, Grimshaw J, Desveaux L, Heisey R, Taccone MS, Taljaard M, Thavorn K, Hodgson D, Gupta S, Lofters A, Ivers N, Nathan PC. Protocol for the ONLOOP trial: pragmatic randomized trial evaluating a province-wide system of personalized reminders for evidence-based surveillance tests in adult survivors of childhood cancer in Ontario. Implement Sci. 2024 Feb 23;19(1):19. doi: 10.1186/s13012-024-01347-x. PMID 38395903